CLINICAL TRIAL: NCT01755754
Title: A Multicenter, Open-label, Randomized, Two-period, Crossover Non-inferiority Trial to Assess the Functionality of Female Condoms With a Silicone Elastomer Vaginal Ring
Brief Title: A Trial to Assess the Functionality of Female Condom With a Silicone Elastomer Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IPM 033
Record Dates: First submitted 2012-12-14; First posted 2012-12-24 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Single-Use Internal Condom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Silicone Elastomer Vaginal Ring (Experimental): Silicone Elastomer Vaginal Ring
  Interventions: Combination Product: Silicone Elastomer Vaginal Ring
- Female Condom (Experimental): This trial will test the performance of female condoms when used concurrently with a placebo vaginal ring
  Interventions: Combination Product: Silicone Elastomer Vaginal Ring; Device: Female Condom

INTERVENTIONS:
Combination Product: Silicone Elastomer Vaginal Ring — Silicone Elastomer Vaginal Ring
Device: Female Condom — Female condom
  Arms: Female Condom

SUMMARY:
A multi-center, open-label, randomized, two-period, crossover non-inferiority trial to assess the functionality of female condoms with a silicone elastomer vaginal ring.

DETAILED DESCRIPTION:
This was an open-label, randomized, 2-period, crossover non-inferiority trial, conducted over 4.5 months at two research centers in the USA among 81 healthy, monogamous, heterosexual, sexually active couples to assess the functionality of female lubricated, nitrile condoms during vaginal intercourse in the presence and absence of a silicone elastomer placebo vaginal ring.

ELIGIBILITY:
Inclusion Criteria:

1. Mutually monogamous heterosexual couples; current relationship ≥3 months; and who can give written informed consent;
2. Age ≥18 to ≤45 years (females) or ≥18 to ≤55 years (males) at time of the screening visit;
3. Healthy on the basis of medical history;
4. Not at risk of pregnancy, i.e., female is surgically sterile, using an IUD, or using effective hormonal contraception, or has a vasectomized partner. The use of vaginal contraceptive rings will not be allowed;
5. Sexually active and agree to have at least 8 acts of penile-vaginal intercourse using a study condom over 2 periods of up to 4 weeks each;
6. Agree to use only the female condoms provided by trial personnel during the time of participation and not to use male condoms during the trial. Additional lubricant will be provided; use of non-study lubricants will not be allowed;
7. Agree to not use genital jewelry or other vaginal products, except menstrual absorption products (e.g., tampons) and study lubricant during the trial;
8. Available for all visits and consent to follow all procedures scheduled for the trial;
9. At low risk for HIV infection.

Exclusion Criteria:

1. Males with untreated erectile dysfunction;
2. Female with positive pregnancy test;
3. Either partner allergic or hypersensitive to vaginal lubricants such as Astorlige ®
4. Either partner not willing to refrain from wearing genital piercing jewelry for the duration of the study
5. History by self-report of recurrent or a recently-treated (within past 2 weeks) sexually transmitted infection (e.g. gonorrhea, syphilis, chlamydia) or HIV(+);
6. Consistently using male or female condoms for protection against sexually transmitted infection;
7. Either partner taking any topical or oral medication to treat a urogenital condition at enrollment, except medication for the male partner to treat erectile dysfunction (e.g., tadalafil, sildenafil);
8. Either partner with a self-reported or clinically diagnosed urogenital condition (e.g. itching, burning, irritation, etc.) that, in the opinion of the Investigator, could affect use of the study condoms or ability to interpret trial data;
9. Females, based on findings from a pelvic examination, who are not suitable candidates for wearing the vaginal ring (anatomical condition, current vaginal infection, etc.)
10. Current participation in a study or other research involving a drug, device or other product;
11. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Total clinical failure rate | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- California Family Health Council, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No